CLINICAL TRIAL: NCT02253446
Title: A Comparison of Analgesic İmpacts of Piroxicam and Diclofenac Sodium in the Treatment of Primary Dysmenorrhea:A Double-Blind, Randomized Trial
Brief Title: A Comparison of Analgesic İmpacts of Piroxicam and Diclofenac Sodium in the Treatment of Primary Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bulent Erdur, professor, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MDhayri2014
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Piroxicam; Diclofenac Sodium; Emergency department
MeSH Terms: conditions — Dysmenorrhea; Emergencies | interventions — Piroxicam; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piroksikam (Experimental): 20 mg of piroxicam (feldene ampoule -Pfizer-France) intramuscularly (IM) was given 200 patients,
  Interventions: Drug: Piroxicam
- Diclofenac Sodium (Experimental): Second Group: Diclofenac sodium 75mg (Miyadren drug-ampoule -Yavuz Istanbul) intramuscularly (IM) was given 200 patients.
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Piroxicam — 20 mg of piroxicam (Feldene ampoule-Pfizer-France) intramuscularly (IM) was given 200 patients,
  Other Names: Feldene 20 mg/1 mL Solution injectable IM
  Arms: Piroksikam
Drug: Diclofenac Sodium — Second Group: Diclofenac sodium 75mg (Miyadren ampoule-bulb-Yavuz Istanbul) intramuscularly (IM) was given 200 patients.
  Other Names: DICLOMEC (Solution injectable IM); DIKLORON (Solution injectable IM ); MIYADREN (Solution injectable IM ); VOLTAREN (Solution injectable IM )
  Arms: Diclofenac Sodium

SUMMARY:
* Currently, nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of patients with Primary Dysmenorrhea.
* The objective of the study is compare intramuscular Diclofenac sodium and piroxicam's pain reduction dysmenorrhea in emergency department (ED) adults.
* The investigators second aim was to compare recurrent dysmenorrhea pain within 24 hours after discharge.

DETAILED DESCRIPTION:
* this is the randomized double blinded clinical trial to compare the efficacy of these two drugs in this clinical setting.
* A randomized clinical trial was conducted in the ED of Pamukkale University Medical Faculty Hospital
* Study personnel (emergency physicians and nurses) were trained before the study.
* When intramuscular drugs (Piroxicam, Diclofenac sodium) was being recommended, an eligibility checklist was completed by the attending physician.
* If there were no exclusion criteria, written informed consent was obtained and baseline information, including initial Dysmenorrhea pain severity ratings with VAS were recorded.
* The need for identification and enrollment of participants by staff with conflicting work pressures resulted in recruitment of a convenience sample of patients.
* All patients eligible for the study were randomized to one of two groups:
* First Group: 20 mg of piroxicam (feldene ampoule -Pfizer-France) intramuscularly (IM) was given 200 patients,
* Second Group: Diclofenac sodium 75mg (Miyadren drug-ampoule -Yavuz Istanbul) intramuscularly (IM) was given 200 patients which determined to be applied as a group.
* Drug packs prepared in 5 ml syringes were numbered by an independent nurse, who not involved in the study.
* Drugs were prepared according to the computer-generated random number sequence to assign treatment allocations
* The allocation list was kept by the emergency nurse. Patients received the piroxicam, diclofenac sodium medication schemes according to their random allocations.
* After enrollment and recording of baseline information, the next numbered study drug pack was obtained, and administered as a intramuscular.
* Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms)
* One researcher blinded to patient allocation observed the whole procedure and recorded the Dysmenorrhea pain scores.
* Patients in both groups received two types of medication in a similar manner, thus ensuring double blinding.
* Dysmenorrhea pain scores were recorded at 0, 15, 30, 45 and 60 min on a VAS of 1 to 10
* Rescue medication (100 mg of tramadol hydrochloride) was given intramuscular to patients if pain VAS scores ≥ 5 in forty five minutes after study drug administration.
* All other medications required during the study also were recorded.
* During the study, pulse rate, systolic blood pressure, diastolic blood pressure, respiration rate and oxygen saturation (SpO2) were recorded at baseline (0 min), 15, 30, and 60 min.

ELIGIBILITY:
Inclusion Criteria:

* patients were eligible for inclusion if they were aged 18 years or older, 45 years or younger
* had Primary Dysmenorrhea
* VAS (visual analog scale) score >5.

Exclusion Criteria:

* Patients with severe liver, kidney and heart failure
* After the use of aspirin or other nonsteroidal antiinflammatory drugs, asthma, nasal polyps, angioedema and urticaria to be seen
* To have active peptic ulcer bleeding or perforation
* Have a history of upper gastrointestinal disease
* The presence of Phenylketonuria disease
* To be Pregnancy and breast-feeding
* To be Asthma patients
* Have received analgesics in the last 4 hours
* Patients of childbearing age who are not using a birth control method.
* The patient who using digoxin, lithium, furosemide and other diuretics, acetylsalicylic acid and anticoagulant coumadin
* Physical examination and suspected acute abdomen.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Compare decrease of dysmenorrhea VAS (visual analog scale) score between the two groups. - (First group Piroxicam and Second Diclofenac Sodium) | Change from Baseline in dysmenorrhea pain VAS scores at 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mehpare camlibel, MD, Principal Investigator — pamukkale universty
Locations (1):
- Pamukkale Universty, Denizli, Denizli, Turkey (Türkiye)